CLINICAL TRIAL: NCT00496366
Title: Phase II Trial of Capecitabine (Xeloda) and Lapatinib (Tykerb) as First-line Therapy in Patients With HER2/Neu-Overexpressing Advanced or Metastatic Breast Cancer
Brief Title: Capecitabine (Xeloda) and Lapatinib (Tykerb) as First-line Therapy in HER2/Neu-positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040608; NJ 1106; 0220070103 (Other: IRB)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer; HER2/Neu-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine (Xeloda) + Lapatinib (Tykerb) (Experimental): Capecitabine for 2 weeks straight (Days 1-14) followed by 1 week without capecitabine (Days 15-21).
  Lapatinib will be taken daily continuously for 21 days (Days 1- 21).
  Interventions: Drug: Capecitabine; Drug: Lapatinib

INTERVENTIONS:
Drug: Capecitabine — The dose of capecitabine is 1000 mg/m2/dose twice each day, orally, 12 hours apart, for 14 consecutive days, every 21 days (total daily dose = 2000 mg/m2).
  Other Names: Xeloda
Drug: Lapatinib — The daily dose of lapatinib is 1250 mg (5 tablets of 250 mg each) to be taken at approximately the same time each day, continuously. Lapatinib is taken even during the week that capecitabine is not taken.
  Other Names: Tykerb

SUMMARY:
Subjects with advanced or metastatic (spread to other parts of the body) breast cancer that is HER2/neu-positive will take part in this study. This type of breast cancer has a high amount of a protein called HER2. HER2 is part of a family of receptors found on both cancer and normal cells. This family of receptors is important for cell growth and is found in many tumor types. The purpose of this research study is to compare an approved treatment for breast cancer capecitabine, also called Xeloda®, to the combination of capecitabine plus an experimental drug, lapatinib also known as Tykerb®, for treatment of advanced or metastatic breast cancer that is HER2/neu-positive.Capecitabine is an approved type of chemotherapy used to treat certain cancers including breast cancer. Capecitabine fights cancer by interfering with the ability of cells to divide and tumor growth. Lapatinib (Tykerb®) is considered "investigational", which means the drug has not been approved by the US Food and Drug Administration (FDA) for sale as a prescription or over-the-counter medication. Lapatinib may slow or stop cancer cells from growing by inhibiting the growth of cancer cells. However, this theory has not been proven. The addition of the study drug (lapatinib) to capecitabine may help stop cancer cells as well as or better than capecitabine alone. Other studies have demonstrated activity and tolerability of lapatinib either alone or in combination with capecitabine in the treatment of breast cancer.Subjects will receive capecitabine and lapatinib. A treatment period will be 21 days long. This period is known as a "cycle". All medications will be given by mouth. Subjects will take capecitabine for 2 weeks straight (Day 1-14) followed by a 1 week without capecitabine (Day 15-21). Doses of lapatinib will be taken daily continuously for 21 days (Day 1-Day 21) which means that subjects will still take lapatinib on the week that they do not take capecitabine (Day 15-21). Subjects will continue to receive these medications unless they experience severe, serious and/or excessive side effects, the cancer becomes worse, the subjects wishes to no longer participate or the study doctor feels it is not in the best interest to continue treatment.Tests and procedures such as physical exam, blood tests, CT or MRI, ECG, ECHO and/or MUGA tests will be conducted at one or more of the following time points: before the study starts, before each cycle, every 6 and 12 weeks, and after the last dose of capecitabine/lapatinib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer
* Stage IIIB, IIIC with T4 lesion or Stage IV disease
* Breast cancer must be determined to be HER2-positive. Assays using fluorescence in situ hybridization (FISH) require gene amplification and assays using immunohistochemistry require a strongly positive (3+) staining intensity score in primary or metastatic tumor tissue
* Measurable disease according to RECIST (Response Evaluation Criteria In Solid Tumors)
* Age ³ 18 years of age
* ECOG performance status 0, 1 or 2 (Appendix B)
* Life expectancy of 3 months or longer
* Able to swallow oral medication
* Adequate end organ function
* Left ventricular ejection fraction
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation
* Written informed consent

Exclusion Criteria:

* Prior treatment with chemotherapy for advanced or metastatic breast cancer
* Prior anti-ErbB1 and/or ErbB2 inhibitor therapy for breast cancer; neoadjuvant or adjuvant treatment with trastuzumab will be allowed provided the last dose was > 6 months prior to enrollment in study
* Symptomatic or untreated brain metastases or carcinomatous meningitis
* Uncontrolled illnesses including symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia requiring therapy, myocardial infarction within the past 6 months, or active infection
* History of other primary malignancies in the last 5 years prior to on-study date except carcinoma in situ of the cervix and nonmelanoma skin cancer
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to capecitabine and/or lapatinib
* Concurrent treatment with other investigational or commercial anti-cancer agent(s)
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Less than 3 weeks since prior radiotherapy
* Less than 2 weeks since prior hormonal therapy
* Known HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with lapatinib
* Pregnant or lactating women at anytime during the study
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Certain medications that act through the CYP450 system are specifically prohibited in patients receiving lapatinib because in vitro data indicate that the agents has the potential to interact with cytochrome P450 enzymes CYP3A4. Certain other agents should be used with caution. Medications that are specifically prohibited can be found in Appendix C.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-07-23 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2017-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Toppmeyer, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We are reporting results on 11 subjects enrolled, who were recruited from July 2007 through December 2009. Subjects were recruited through the Cancer Institute of New Jersey's Oncology Group and this study was closed pre-maturely due to slow accrual.
Groups:
- Capecitabine (Xeloda) + Lapatinib (Tykerb): Capecitabine for 2 weeks straight (Days 1-14) followed by 1 week without capecitabine (Days 15-21).
  Lapatinib will be taken daily continuously for 21 days (Days 1- 21).
  Capecitabine: The dose of capecitabine is 1000 mg/m2/dose twice each day, orally, 12 hours apart, for 14 consecutive days, every 21 days (total daily dose = 2000 mg/m2).
  Lapatinib: The daily dose of lapatinib is 1250 mg (5 tablets of 250 mg each) to be taken at approximately the same time each day, continuously. Lapatinib is taken even during the week that capecitabine is not taken.
Period: Overall Study
Arm/Group | Capecitabine (Xeloda) + Lapatinib (Tykerb)
Started | 11
Completed | 10
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine (Xeloda) + Lapatinib (Tykerb)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 60.7 [39 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Determine the Response Rate (as Determined by RECIST Criteria) of Capecitabine and Lapatinib as First-line Therapy in Patients With Advanced or Metastatic Breast Cancer That Overexpress HER2.
Time Frame: 2 years
Population: Study to was terminated early and insufficient data was collected to assess this outcome measure.
Arm/Group | Capecitabine (Xeloda) + Lapatinib (Tykerb)
Number analyzed (Participants) | 0
Value | 0

2. Secondary Outcome: -Determine the Clinical Benefit Rate (Complete Response, Partial Response, or Stable Disease for at Least 6 Months) of Capecitabine and Lapatinib. -Determine Time to Disease Progression After Treatment With Capecitabine and Lapatinib. -Evaluate Overall
Time Frame: 2 years
Population: Study was terminated early and insufficient data was collected to assess this outcome measure.
Arm/Group | Capecitabine (Xeloda) + Lapatinib (Tykerb)
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Arm/Group | Capecitabine (Xeloda) + Lapatinib (Tykerb)
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine (Xeloda) + Lapatinib (Tykerb) (N=11)
Sepsis (Infections and infestations) | 1 (1)
Death (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine (Xeloda) + Lapatinib (Tykerb) (N=11)
Fatigue (General disorders) | 4 (9)
Weight loss (Investigations) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 6 (19)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 5 (11)
Dysgeusia (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8)
Vomiting (Gastrointestinal disorders) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Mucositis - oral (Gastrointestinal disorders) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophiles (Infections and infestations) | 2 (4)
Infection with unknown ANC (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes